CLINICAL TRIAL: NCT04474431
Title: Correlation of VEGF-A and Fluid Balance in Septic Shock
Acronym: VEGFluid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018/0346/HP
Record Dates: First submitted 2020-06-25; First posted 2020-07-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients admitted in the ICU of hospital of Rouen (Other): Patients admitted in the intensive care unit (ICU) of the teaching hospital of Rouen.
  Interventions: Other: Evaluation of VEGF-A levels in patients with septic shock is positively correlated with a positive fluid balance.

INTERVENTIONS:
Other: Evaluation of VEGF-A levels in patients with septic shock is positively correlated with a positive fluid balance. — Evaluation of VEGF-A levels in patients with septic shock is positively correlated with a positive fluid balance.

SUMMARY:
VEGF is a key molecule in the control of vascular permeability via interactions with the VEGF-receptor on the endothelial cell. Several authors reported plasma VEGF levels are elevated in sepsis shock and associated with increased mortality (1,2).

In septic shock, the main elements of treatment are intravenous fluids, appropriate antibiotics and vasopressors. Some authors observed positive fluid balance is associated with increased mortality rates in patients (3,4).

To the best of our knowledge, no studies have shown a correlation between VEGF levels and the fluid balance. The aim of our study was to determine the role of VEGF in capillary leakage and the positive fluid balance in septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18 years old
* Patient with septic shock (presence of an infection, hypotension with mean arterial pressure less than 65mmHg and the need for vasopressor treatment (minimum dose 0,3µ/kg/min)
* Person informed and signed consent.

Exclusion Criteria:

* Death predicted within 24 hours
* Limitation of therapeutic attitudes
* Treatment with bevacizumab in the past 6 months
* Pathologies with endothelial dysfunction (scleroderma, clarkson syndrome...)
* Acute renal failure (KDIGO 3) at ICU admission defined by :
* Increase in serum creatinine to > 354µmol/l or 3 times baseline OR
* Urine output ≤0,3 ml/kg/h for 24h OR
* Anuria for 12h
* Morbid obesity with a body mass index (BMI) > 35 kg/m².
* Limb amputation
* Morbid obesity with a body mass index (BMI) > 35 kg/m².
* Amputation of a limb
* Pregnant or nursing women
* Inability to obtain consent from family
* Person with guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Show that elevation of VEGF-A levels at D1 in the management of patients with septic shock is positively correlated with a positive fluid balance. | 1 day
  Plasma assay of the VEGF-A by enzyme-linked immunosorbent assay (ELISA) and calculated fluid balance at D1 of ICU admission.

SECONDARY OUTCOMES:
Correlation of VEGF-A levels and fluid balance at D3 of ICU admission. | 3 days
  Plasma assay of the VEGF-A by enzyme-linked immunosorbent assay (ELISA) and calculated fluid balance at D3 of ICU admission.
Correlation of VEGF-A levels with edema at D1 and D3 of ICU admission. | 1 and 3 days
  Plasma determination of endothelial dysfunction biomarkers by the enzyme-linked immunosorbent assay (ELISA) method: VEGF-A at D1 and D3 of ICU admission edema evaluation at D1 and D3 of ICU admission by:
  * Weight
  * fluid balance: difference between input (fluid therapy) and output (urine output)
  * Ultrasound-measured thickness of subcutaneous tissue
  * Measurement of total, intra and extra cellular body water evaluated by bioimpedancemetry
Correlation of Soluble Vascular Endothelial Growth Factor Receptor 1 (sFlt1) levels and edema at D1 and D3 of ICU admission. | 1 and 3 days
  Plasma determination of endothelial dysfunction biomarkers by the enzyme-linked immunosorbent assay (ELISA) method: sFlt1 at D1 and D3 of ICU admission edema evaluation at D1 and D3 of ICU admission by:
  * Weight
  * fluid balance: difference between input (fluid therapy) and output (urine output)
  * Ultrasound-measured thickness of subcutaneous tissue
  * Measurement of total, intra and extra cellular body water evaluated by bioimpedancemetry
Correlation of sFlt1 levels and fluid balance at D1 and D3 of ICU admission. | 1 and 3 days
  Plasma determination of endothelial dysfunction biomarkers by the enzyme-linked immunosorbent assay (ELISA) method: sFlt1
  - fluid balance: difference between input (fluid therapy) and output (urine output)
Correlation of VEGF A levels and microcirculation at D1 and D3 of ICU | 1 and 3 days
  Plasma determination of endothelial dysfunction biomarkers by the enzyme-linked immunosorbent assay (ELISA) method: VEGF-A Study of microcirculation in vivo by Glycocheck: capillary density, Blood flow and red cell velocity, Endothelial glycocalyx function at D1 and D3 of ICU admission
Evolution of VEGF A and sFLT1 levels between D1 and D3 of ICU admission. | 1 and 3 days
  Plasma determination of endothelial dysfunction biomarkers by the enzyme-linked immunosorbent assay (ELISA) method: VEGF-A and sFlt1 at D1 and D3 of their management in intensive care units.
Correlation of VEGF A levels at D1 and mortality at D28 of management. | 28 days
  Survival at D28 of ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rouen, Rouen, France